CLINICAL TRIAL: NCT06335706
Title: The Influence of Fit of Underpants Worn on Semen Quality
Status: Completed | Type: Observational
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Harnam Kaur, MD, Principal Investigator, Chulalongkorn University
Other Study IDs: 0596/66
Record Dates: First submitted 2024-03-14; First posted 2024-03-28 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Infertility, Male; Semen Analysis
Keywords: Fit of underpants worn; Genital heat stress; Basic semen parameters; Sperm DNA integrity; Thai male partners
MeSH Terms: conditions — Infertility, Male

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frequently worn underpants during daytime: It will be divided into two groups based on the type of underwear worn: loose-fit, which includes boxers and tight-fit, which includes all other types.
  Interventions: Behavioral: Fit of underpants worn
- Frequently worn underpants at nighttime: It will be divided into two groups based on the type of underwear worn: loose-fit, which includes boxers or none, and tight-fit, which includes all other types.
  Interventions: Behavioral: Fit of underpants worn

INTERVENTIONS:
Behavioral: Fit of underpants worn — Tight or loose-fitted underpants

SUMMARY:
The goal of this observational study is to investigate the impact of underpants fit among Thai males attending the Infertility Clinic, whether alone or with their spouses. The main questions it aims to answer are:

* Assessing the effect of underpants fit on basic semen parameters and sperm DNA integrity.
* Determining the prevalence of preferred type of underpants worn by Thai males.

The participants will need to provide informed consent, complete a questionnaire consisting of 28 questions, and provide a semen sample.

DETAILED DESCRIPTION:
This research aims to investigate the impact of underpants fit on basic semen parameters, with secondary objectives including an examination of its effect on sperm DNA integrity and an assessment of the prevalence of different underpants types among Thai male partners. The study will enroll approximately 120 Thai male partners, aged 20-55 years, attending the Reproductive Biology Unit (Infertility Clinic) at King Chulalongkorn Memorial Hospital in Bangkok, Thailand, either alone or with their spouses. Participants will be required to provide informed consent, complete a 28-question questionnaire, which should take no more than 10 minutes, and undergo semen analysis. The analysis will assess basic semen parameters and sperm DNA integrity, preferably after a 2-7 days abstinence period. The research will be conducted over a single day for each participant.

The data will be divided into two groups based on underpants fit: loosely fitted and tightly fitted. Statistical analysis will be conducted using STATA software version 18, employing regression analysis to assess the independent impact of underpants fit on semen quality. This analysis will control for potential confounding factors such as age, obesity, alcohol and caffeine consumption, cigarette smoking, physical activity, excessive heat exposure, recreational drug use, recent COVID-19 infection, duration of abstinence, previous children, and stress.

This study seeks to build on previous findings, address genital heat stress in Thai male partners, and potentially influence lifestyle changes to reduce male-factor infertility. Future research could explore additional factors such as underwear material and the type of trousers worn by men.

ELIGIBILITY:
Inclusion Criteria:

* Male partner, Thai citizen
* Age 20 - 55 years
* Participants able and willing to fill in an informed consent form
* Participants capable of completing questionnaire form
* Semen sample collection after 2-7 days of abstinence
* Participants wearing specific type of underpants not less than 8 hours per day

Exclusion Criteria:

* Any congenital factor (e.g. cystic fibrosis, congenital absence of vas deferens, cryptorchidism)
* Any testicular disorder (e.g. varicocele, testicular torsion, testicular trauma)
* Any genital tract disorders/ infections (e.g. prostatitis, epididymitis, urogenital tract obstruction)
* Severe systemic disorder (e.g. liver cirrhosis, renal failure)
* Sexual dysfunction (erectile dysfunction)
* Exogenous factors (chemotherapy, medications, radiation)
* Any surgery comprising vascularization of testis
* Participants wearing both tight and loose-fitted underpants

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender: Male Eligibility Criteria: Male individuals, aged 20-55 years, and citizens of Thailand.
Study Population: The study aims to enroll approximately 120 participants, comprising Thai male partners who either alone or with spouses visit the Reproductive Biology Unit (Infertility Clinic) at King Chulalongkorn Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-03-28 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Semen Volume | Semen sample will be collected once, on a date advised by the doctor, following a period of ejaculatory abstinence ranging from 2 to 7 days. The sample will be evaluated within 30 minutes of collection.
  Semen volume will be assessed in milliliters.
Total sperm count | Semen sample will be collected once, on a date advised by the doctor, following a period of ejaculatory abstinence ranging from 2 to 7 days. The sample will be evaluated within 30 minutes of collection.
  The total sperm count will be assessed as the total number of sperm cells in millions in the entire ejaculate.
Sperm concentration | Semen sample will be collected once, on a date advised by the doctor, following a period of ejaculatory abstinence ranging from 2 to 7 days. The sample will be evaluated within 30 minutes of collection.
  Sperm concentration will be quantified as the number of million sperm cells per milliliter.
Sperm motility | Semen sample will be collected once, on a date advised by the doctor, following a period of ejaculatory abstinence ranging from 2 to 7 days. The sample will be evaluated within 30 minutes of collection.
  Sperm motility will be evaluated as the percentage of sperm cells exhibiting movement.
Sperm morphology | Semen sample will be collected once, on a date advised by the doctor, following a period of ejaculatory abstinence ranging from 2 to 7 days. The sample will be evaluated within 30 minutes of collection.
  Sperm morphology will be evaluated as percentage of sperm cells with normal shape.

SECONDARY OUTCOMES:
Sperm DNA integrity | The leftover semen sample after basic semen analysis will be stored and slides will be prepared. Sperm DNA integrity will be assessed immediately after slide preparation or after freezing the slide for one day, if necessary.
  Sperm DNA integrity will be evaluated as percentage of abnormal DNA fragmentation (%).

OTHER OUTCOMES:
Preferred type of underpants | The analysis will commence upon completion of the anticipated data collection period of 3-months.
  It will be evaluated as the percentage of participants who predominantly wear different types of underwear.

CONTACTS AND LOCATIONS:
Overall Officials: Unnop Jaisamrarn, MD, MHS, Study Chair — Chulalongkorn University; Harnam Kaur, MBBS, Principal Investigator — Chulalongkorn University
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Undecided